CLINICAL TRIAL: NCT04728542
Title: A Post-market Observational ORIGIN® vs. VANGUARD® PS Clinical Study: a Comparative, Prospective, Randomized Controlled Clinical and Radiological Evaluation.
Brief Title: ORIGIN® vs. VANGUARD® PS Observational Study
Status: Recruiting | Type: Observational
Sponsor: Symbios Orthopedie SA (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-G-010; 2019-14580 (Other: Landersarztekammer Rheinland-Pfal)
Record Dates: First submitted 2021-01-20; First posted 2021-01-28 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Arthroplasty; Replacement; Knee
Keywords: Arthroplasty; Knee; Prosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Origine: 70 subjects with the ORIGIN PS System
  Interventions: Device: ORIGIN PS System
- Vanguard: 70 subjects with the VANGUARD System
  Interventions: Device: VANGUARD PS System

INTERVENTIONS:
Device: ORIGIN PS System — 70 surgeries with the ORIGIN PS System
  Groups: Origine
Device: VANGUARD PS System — 70 surgeries with the VANGUARD System
  Groups: Vanguard

SUMMARY:
The study objective is to assess patient satisfaction after the surgery with a patient match CE marked implant (ORIGIN®) versus off-the-shelf (VANGUARD PS) device, and to document the clinical and device performance outcomes of the ORIGIN System used in routine hospital practice in a large patient cohort treatment of total knee arthroplasty.

DETAILED DESCRIPTION:
This is a prospective, comparative, randomized, double arm, monocentric, observational, post-market study with 140 subjects with 2 years follow-up.

ELIGIBILITY:
Inclusion/exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-inflammatory degenerative and inflammatory knee joint disease
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Forgotten Joint Score | Preoperative, 1 year, and 2 years visits
  12 questions and measure the ability of the patient to forget their operated knee after the surgery.
The Self-Administered Patient Satisfaction Scale | Preoperative, 1 year, and 2 years visits
  Patients' overall satisfaction with surgery, the extent of pain relief, the ability to perform home or yard work, and the ability to perform recreational activities.

SECONDARY OUTCOMES:
Oxford Knee Score (OKS) | Preoperative, 1 year, and 2 years visits
  Patient reported scores This Quality of Life score was developed in 1998 and validated to measure pain and function after total knee replacement. It consists of 12 questions about pain, function and mobility of the knee joint.
  Each question scores from 1 to 5 (1 the best and 5 the worst) and the sum of all the scores is deducted from 60 points. The best total is 48 points and the worst is 0.
EQ-5D-5L | Preoperative, 1 year, and 2 years visits
  Patient reported scores.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can image' and 'The worst health you can image'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Knee Society clinical rating system (KSS) Objective Knee Indicators | Preoperative, 1 year, and 2 years visits
  Surgeon reported score.
  It consists of 4 questions regarding the alignment and mobility of the knee joint:
  "Alignment" has a maximum of 25 points and is determined on a weight-bearing AP radiograph measuring the femoral-tibial (Anatomic) axis.
  "Instability" allows a maximum of 25 points for a knee that is stable in the coronal and saggital axis.
  "Joint Motion" allows one point for each 5° of joint motion. Unlike the old scoring system that allowed a maximum of 25 points the new system allows greater than 25 points for patients with greater than 125° of motion. There are deductions for flexion contracture and extension lag. The presence of recurvatum is not specifically addressed however patients with recurvatum will have significant ligament laxity in other planes that is captured in the
  "Instability" category of the objective score. Maximum allowable points 25+
Single Leg Stance test | Preoperative, 1 year, and 2 years visits
  Surgeon reported score. It is used to assess static postural and balance control. It is a balance assessement that is widely used in clinical settings to monitor neurological and musculoskeletal conditions.
  It measures the duration of exercices with eyes opened and closed in seconds.
Time Up & Go tests | Preoperative, 1 year, and 2 years visits
  Surgeon reported score It is a simple test to assess a person's mobility and requires both static and dynamic balance (e.g. Getting up from a chair with armrests, Make a U turn...) The criteria are : able - unable

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Drees, Prof, Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- University Medical Center of Johannes Gutenberg-University Mainz, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlson VR, Post ZD, Orozco FR, Davis DM, Lutz RW, Ong AC. When Does the Knee Feel Normal Again: A Cross-Sectional Study Assessing the Forgotten Joint Score in Patients After Total Knee Arthroplasty. J Arthroplasty. 2018 Mar;33(3):700-703. doi: 10.1016/j.arth.2017.09.063. Epub 2017 Oct 7. PMID 29108793
- [Background] Wheatley B, Nappo K, Fisch J, Rego L, Shay M, Cannova C. Early outcomes of patient-specific posterior stabilized total knee arthroplasty implants. J Orthop. 2018 Dec 6;16(1):14-18. doi: 10.1016/j.jor.2018.11.003. eCollection 2019 Jan-Feb. PMID 30765928
- [Background] Kahlenberg CA, Lyman S, Joseph AD, Chiu YF, Padgett DE. Comparison of patient-reported outcomes based on implant brand in total knee arthroplasty: a prospective cohort study. Bone Joint J. 2019 Jul;101-B(7_Supple_C):48-54. doi: 10.1302/0301-620X.101B7.BJJ-2018-1382.R1. PMID 31256639